CLINICAL TRIAL: NCT07253337
Title: Effect of First Premolars Extraction During Orthodontic Treatment on Distribution of Bite Force During the Mandibular Excursive Movements: A Prospective Clinical Trial Using T-scan Occlusal Analysis System.
Brief Title: Analysis of Bite Force Distribution After Premolars Extraction by Using T-scan Analysis System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, rim fathalla, Rim Mohamed Fathalla Eissa, Suez Canal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1041/2025
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Effect of Premolars Extraction on Bite Force
Keywords: occlusion T-scan extraction

STUDY DESIGN:
Intervention Model Description: T-scan analysis for distribution of bite force before and after the end of the orthodontic treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with premoalrs extraction (Experimental): Patients who will undergo 4 first premolars extraction Patients who will undergo upper first premolars extraction
  Interventions: Other: T-scan analysis for bite force distribution

INTERVENTIONS:
Other: T-scan analysis for bite force distribution — T-scan analysis for bite force distribution for patients before and after the end of the orthodontic treatment

SUMMARY:
This study aims to assess the effect of first premolars extraction during orthodontic treatment bite force during the excursive mandibular movements using a digital occlusal analysis system.

DETAILED DESCRIPTION:
The study sample consists of 16 patients, aged 14-25 years-old, who will be presented at the outpatient dental clinics and are seeking orthodontic treatment to relief crowding or to treat their proclined teeth. A written consent will be signed by them or their parents or caregivers after their approval to participate in this research study. The inclusion criteria are : age group from14 to 25 years, full complement of permanent teeth (excluding third molars) and the case analysis revealed extraction of their first premolars to relieve the malocclusion problem. As for the exclusion criteria; they include patients with previous Orthodontic/ Orthopedic/ Orthognathic surgical treatment, patients with history of trauma or obvious/ gross facial asymmetry.

Patients sampling:

Patients will be divided into two groups , each group includes eight patients according to the proposed treatment plan:

* Group I : Patients who will be treated with the extraction of their upper and lower first premolars .
* Group II : Patients who will be treated with extraction of their upper first premolars.

Methods:

Records will be taken on patients selected before initiating any orthodontic treatment to register the occlusal force distribution on teeth during the different excursive mandibular movements (right, left and protrusive mandibular movements) using the T-scan III system before orthodontic treatment and extraction of teeth .

* Orthodontic treatment of patients will be undertaken.
* After finishing the patients' treatment , the T-scan III system is used to measure the bite force distribution during mandibular excursive movements immediately after brackets debonding .
* The bite force measurements taken before and after treatment will be compared with each other .

Statistical Analysis:

In the current study, observations and all numerical data will be collected for statistical analysis using SPSS version 29 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Age group from14 to 25 years
* Full complement of permanent teeth (excluding third molars)
* The case analysis revealed extraction of their first premolars to relieve the malocclusion problem

Exclusion Criteria:

* Patients with previous Orthodontic/ Orthopedic/ Orthognathic surgical treatment
* Patients with history of trauma or obvious/ gross facial asymmetry.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of bite force during excursive mandibular movements | 12-18 months
  Distribution of bite force during excursive mandibular movements before and after the end of the orthodontic treatment

SECONDARY OUTCOMES:
Effect of premolars extraction on distribution of bite force during mandibular excursive movements | 12-18 months
  Effect of first premolars extraction on distribution of bite force during mandibular excursive movements using T-scan occlusal analysis system and if the extraction pattern is acontributing factor in the bite force

CONTACTS AND LOCATIONS:
Overall Officials: Rim M Fathalla, PhD of Orthodontics, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sultana MH, Yamada K, Hanada K. Changes in occlusal force and occlusal contact area after active orthodontic treatment: a pilot study using pressure-sensitive sheets. J Oral Rehabil. 2002 May;29(5):484-91. doi: 10.1046/j.1365-2842.2002.00849.x. PMID 12028498
- [Result] Bottger H, Borgstedt T. [Computer-supported analysis of occlusion using T-Scan system. First report]. ZWR. 1989 Jul;98(7):584-5. German. PMID 2700857
- [Result] Floystrand F, Kleven E, Oilo G. A novel miniature bite force recorder and its clinical application. Acta Odontol Scand. 1982;40(4):209-14. doi: 10.3109/00016358209019814. PMID 6958166
- [Result] Helkimo E, Carlsson GE, Helkimo M. Bite force and state of dentition. Acta Odontol Scand. 1977;35(6):297-303. doi: 10.3109/00016357709064128. PMID 271452
- [Result] Rohrle O, Saini H, Ackland DC. Occlusal loading during biting from an experimental and simulation point of view. Dent Mater. 2018 Jan;34(1):58-68. doi: 10.1016/j.dental.2017.09.005. Epub 2017 Oct 7. PMID 29017762
- [Result] Sharma A, Rahul GR, Poduval ST, Shetty K, Gupta B, Rajora V. History of materials used for recording static and dynamic occlusal contact marks: a literature review. J Clin Exp Dent. 2013 Feb 1;5(1):e48-53. doi: 10.4317/jced.50680. eCollection 2013 Feb 1. PMID 24455051
- [Result] Haydar B, Ciger S, Saatci P. Occlusal contact changes after the active phase of orthodontic treatment. Am J Orthod Dentofacial Orthop. 1992 Jul;102(1):22-8. doi: 10.1016/0889-5406(92)70011-x. PMID 1626529